CLINICAL TRIAL: NCT00001662
Title: Tolerability and Primary Efficacy of CX516 in Alzheimer's Disease
Brief Title: Treatment of Alzheimer's Disease With CX516 (Ampalex)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 970049; 97-N-0049; NCT00000181 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-11

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: Dementia; Glutamate; Clinical Trial; Neurotransmitter; Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — 1-(quinoxalin-6-ylcarbonyl)piperidine

INTERVENTIONS:
Drug: CX516 (Ampalex)

SUMMARY:
Glutamate is an amino acid released by brain cells that acts to excite other cells. Glutamate attaches to special sites on cells called AMPA (alpha-amino-2,3-dihydro-5 methyl 3-oxo-4-isoxazolepropanoic acid) receptors. The brain cells responsible for releasing glutamate are damaged in Alzheimer's disease and other conditions affecting thinking and reasoning.

Researchers would like to see if giving patients a drug that attaches to AMPA receptors improves the symptoms of Alzheimer's disease.

CX516 (Ampalex) is a test drug that affects the AMPA receptors. This study will investigate the effectiveness and safety of CX516 on patients with Alzheimer's disease.

Patients will be given capsules of CX516 or placebo (sugar pill that neither harms nor helps) for up to 16 weeks in different amounts. The effectiveness of the drug will be measured by neurological tests. Safety will be monitored by frequent check-ups and lab examinations.

DETAILED DESCRIPTION:
Stimulation of neuronal excitatory amino acid receptors is an important step in the formation of memory. It is unknown whether stimulation of these receptors in patients with Alzheimer's disease and dementing disorders will improve cognitive function. To determine whether positive modulation of AMPA receptors, active in animal models of dementia, can improve cognitive function in demented patients, CX516, at a dose of 900mg TID, will be administered orally for 12 weeks in patients with dementia. In this randomized, controlled proof-of-principle study, drug-induced alterations in intellectual function will be measured by standardized neuropsychological tests. Safety will be monitored by frequent clinical assessments and laboratory tests.

ELIGIBILITY:
INCLUSION CRITERIA - ALZHEIMER'S DISEASE:

Study subjects will satisfy NINCDS-ADRDA criteria for probable Alzheimer's disease.

Dementia severity will be mild to moderate range with Mini-Mental Status Examination total score between 12 and 26, inclusive.

The modified Hachinski Ischemia Score must be less than 4, and brain MRI performed within 15 months of enrollment must be compatible with the diagnosis of Alzheimer's disease.

Dementia must be present historically for at least one year. Baseline electroencephalogram must not show significant epileptiform features.

INCLUSION CRITERIA - RELATED DEMENTING DISORDERS:

Study subjects will show deficits in at least two cognitive spheres, including memory.

Modified Hachinski Ischemia Score must be less than 4, and Folstein mini-mental status examination total score must be between 12 and 26.

Cognitive difficulties must e present historically for at least one year.

Brain MRI performed with 15 months of enrollment must be normal or show atrophy.

Baseline electroencephalogram must not show epileptiform features.

In addition, all patients must have acceptable nutritional status.

Patients must be between ages 40 and 85.

Patients must be sterile, post-menopausal, or using an acceptable forms of birth control.

Chest x-ray within 15 months before enrollment must be acceptable for the trial.

Participants in this study will reflect the diversity of those suffering from dementia.

No one will be excluded or discriminated against based on the grounds of race, creed, or gender.

Every attempt will be made to include women and minorities in the study population.

EXCLUSION CRITERIA - NEUROLOGIC:

Hemispheric stroke, hydrocephalus, subdural hematoma, or mass lesion on neuroimaging study; "epileptiform" baseline EEG or known seizure disorder; head trauma with loss of consciousness concurrent with onset of dementia; chronic CNS infection (positive MHA-TP or FTA-ABS acceptable if luetic brain disease excluded by documented studies or treatment).

EXCLUSION CRITERIA - GENERAL MEDICAL:

Acute serious infection, including hepatitis; hypothyroidism (TSH greater than 6.0 microunits/mL); folic acid deficiency (less than 0.9 ng/mL); vitamin B12 deficiency (less than 160 pg/mL) within one year prior to enrollment; severe renal insufficiency (creatinine clearance less than 25 mL/min, BUN greater than 40 mg/dL, or serum creatinine greater than 2.0 mg/dL); hepatic insufficiency (SGPT or SGOT greater than 3 x upper limit of normal, or total bilirubin greater than 2.0 mg/dL). Due to the serious adverse event transient agranulocytosis report in another study of CX516, patients will neutropenia or low normal white blood cell counts (greater than or equal to 3.5 K/microliter) will be excluded from this study.

PSYCHIATRIC:

Depression if present during screening. Depression will be diagnosed clinically and with depression rating scale(s), such as Hamilton Depression Rating Scale, if needed.

PREVIOUS AND CONCOMITANT MEDICATIONS:

Administration of tacrine, donepezil, rivastigmine, galantamine, anti-depressants are prohibited within thirty days prior to enrollment.

OTHER CONDITIONS:

Any hepatic, cardiovascular, gastrointestinal, or hematological illness which could interfere with drug absorption, distribution, metabolism, or excretion; known hypersensitivity to CX516 or its vehicle; inability to swallow tablets or to comply with medication schedule; no significant care giver; uncorrectable loss of hearing or eyesight that precludes psychometric testing; inability to comprehend instructions or to respond to test items.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 1996-12; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Arai A, Kessler M, Rogers G, Lynch G. Effects of a memory-enhancing drug on DL-alpha-amino-3-hydroxy-5-methyl-4-isoxazolepropionic acid receptor currents and synaptic transmission in hippocampus. J Pharmacol Exp Ther. 1996 Aug;278(2):627-38. PMID 8768713
- [Background] Granger R, Staubli U, Davis M, Perez Y, Nilsson L, Rogers GA, Lynch G. A drug that facilitates glutamatergic transmission reduces exploratory activity and improves performance in a learning-dependent task. Synapse. 1993 Dec;15(4):326-9. doi: 10.1002/syn.890150409. PMID 8153879
- [Background] Greenamyre JT, Maragos WF, Albin RL, Penney JB, Young AB. Glutamate transmission and toxicity in Alzheimer's disease. Prog Neuropsychopharmacol Biol Psychiatry. 1988;12(4):421-30. doi: 10.1016/0278-5846(88)90102-9. PMID 2900537